CLINICAL TRIAL: NCT04212117
Title: Can the Digital Patient Activated Learning System Increase Racial Minority Engagement With Health Information? A Multi-Site Pilot Examination in New York State
Brief Title: CALS Patient Activated Learning System (PALS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 19-08020714
Record Dates: First submitted 2019-12-23; First posted 2019-12-26 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Communication; Trust; Health Knowledge, Attitudes, Practice
MeSH Terms: conditions — Communication; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 - Educational Platform, PALS (Other): The Patient Activated Learning System is a free, health education platform written bu trusted MDs.
  Interventions: Other: The Patient Activated Learning System (PALS)
- Arm 2 - WebMD (Other): WebMD is a widely used educational platform for health information.
  Interventions: Other: WebMD

INTERVENTIONS:
Other: The Patient Activated Learning System (PALS) — Randomization into PALS arm.
  Arms: Arm 1 - Educational Platform, PALS
Other: WebMD — Randomization into WebMD arm.
  Arms: Arm 2 - WebMD

SUMMARY:
The overall goal in this line of inquiry is to test whether the Patient Activated Learning System (PALS) is effective in reducing disparities in access to reliable, easily understood health information, and whether this increased understanding has downstream consequences such as increases in trust in the medical system and self-management behaviors.

DETAILED DESCRIPTION:
Participants will view, in randomized order, PALS or WebMD content on hypertension and on high cholesterol. This study will test knowledge uptake across topics as well as attitudes toward and trust in the information and information providers.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years of age.
* Self-reported hypertension diagnosis.
* English speaking
* Passing the cognition screener
* Able to read in English
* Patient at designated recruitment clinics

Exclusion Criteria:

* Non-English speakers
* Not having self-identified as having hypertension
* Inability to read in English
* Being younger than 18
* Not passing the screener
* Not being a patient on the participating clinics

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Knowledge | Day 1, Immediately after reading article
  as measured by assessment questions on the nutrition information provided
Trust in eHealth | Day 1, Immediately after reading article
  as measured by e-Health Impact Questionnaire by Kelly et al. on a 5-point likert scale where one is strongly disagree and 5 is strongly agree
E-health usability | Day 1, Immediately after reading article
  as measured by e-Health Impact Questionnaire scale by Harris et al. on a 5-point likert scale where one is strongly disagree and 5 is strongly agree
Physician trust | Day 1, Immediately after reading article
  as measured by assessment questions from Wake Forest Physician Trust Scale on a 5-point likert scale where one is strongly disagree and 5 is strongly agree

CONTACTS AND LOCATIONS:
Overall Officials: Neil Lewis, PhD, Principal Investigator — Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No